CLINICAL TRIAL: NCT01548690
Title: A Phase 2a Study to Evaluate the Safety and Tolerability of OCR-002 (Ornithine Phenylacetate) in the Treatment of Patients With Acute Liver Failure/Severe Acute Liver Injury
Brief Title: Safety Study of Ornithine Phenylacetate to Treat Patients With Acute Liver Failure/Severe Acute Liver Injury
Acronym: STOP-ALF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: William Lee (Other)
Collaborators: Medical University of South Carolina (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Ocera Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, William Lee, Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALFSG-OCR-002; U01DK058369 (NIH)
Record Dates: First submitted 2012-02-24; First posted 2012-03-08 (Estimated); Results first posted 2018-09-20 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Acute Liver Failure; Acute Liver Injury
Keywords: ornithine; phenylacetate; acetaminophen toxicity; acute liver failure; hepatitis B; autoimmune hepatitis; drug-induced liver injury
MeSH Terms: conditions — Liver Failure, Acute; Hepatitis B; Hepatitis, Autoimmune; Chemical and Drug Induced Liver Injury | interventions — ornithine phenylacetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ornithine·Phenylacetate (Experimental): Ornithine Phenylacetate is administered intravenously, through a peripheral venous catheter. Each infusion should will be administered over a period of 120 hours.
  Interventions: Drug: Ornithine Phenylacetate

INTERVENTIONS:
Drug: Ornithine Phenylacetate — Up to 36 patients will be enrolled into 2 groups [~18 with minimal renal dysfunction (Cohort 1) & ~18 w/ comprised renal function (Cohort 2)] and receive OCR-002 infusion for at least 72 hrs. OCR-002 will be administered in the vein and pharmacokinetics (pk) assessed for all subjects who receive the infusion.
  The first 24 enrolled subjects received OCR-002 at 3 ascending dose levels (DLs 1-3) with a maximum target infusion rate equivalent to 10g/24h.
  The remaining 12 patients (~6 Cohort 1 & ~6 Cohort 2) will be enrolled and receive identical quantities of OCR-002 at 20g/24hr continuously for 5 days (Dose Level 4).
  Other Names: OCR-002

SUMMARY:
This Phase 2a clinical study is designed to provide data on OCR-002 in patients with acute liver failure/acute liver injury (ALF/ALI) in regard to:

* safety and tolerability;
* metabolism of the compound to glutamine and phenylacetylglutamine (PAGN);
* its effect on circulating ammonia levels and neurological function in patients with and without impaired renal function after continuous infusion at different infusion rates.

Subjects will receive up to 120 hours (5 days) of drug infusion, followed by a 30 day follow-up visit post infusion. It is anticipated that this early safety and tolerability study, with appropriate PK/PD data, will lead to a development program for the use of OCR-002 in the treatment of hyperammonemia either due to ALF or possibly other liver conditions. The hypotheses are:

* Treatment with OCR-002 is safe and tolerable in patients with acute liver failure/acute liver injury due to acetaminophen overdose or drug-induced liver injury, autoimmune hepatitis, viral hepatitis or indeterminate etiologies.
* A dose of 10-20g/24h (0.42-.83g/h) will achieve steady state plasma concentrations within 6-12h with little additional accumulation in the ALI/ALF setting.
* Treatment with OCR-002 will reduce ammonia and improve neurological function in patients with acute liver failure/severe acute liver injury.

DETAILED DESCRIPTION:
There is strong experimental and clinical rationale for the use of ammonia-lowering therapies in ALF. Ammonia is normally produced in the gut and transformed by the liver into urea. As the liver fails, ammonia increases in the systemic circulation and enters into the brain. The result of a rapid rise in ammonia or related compounds in the cerebral circulation is hepatic encephalopathy (HE), a reversible neuropsychiatric condition that ranges in severity from mild impairment in attention, to delirium, the development of cerebral edema, coma and death. This is a Phase 2a, multi-center, open-label study, conducted in two cohorts in patients diagnosed with acute liver failure/acute liver injury (ALF/ALI) who meet inclusion/exclusion criteria. This study is designed to provide data on OCR-002 with regards to

* the effect on circulating ammonia levels in patients with acute liver failure with and without impaired renal function at different doses after single and continuous infusion
* safety and dose tolerability as well as
* providing data on the metabolites, glutamine and phenylacetylglutamine in this patient population.

It is anticipated that this early efficacy, safety, tolerability, Pharmacokinetic/Pharmacodynamic (PK/PD) and dose-ranging study will lead to a Phase 3 development program for the use of OCR-002 in the treatment of hyperammonemia due to ALF. No clinical outcome measures will be formally studied because of the small sample size.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, ages 18-65 (have not reached their 66th birthday).
2. Acute liver failure, defined as the development of coagulopathy (International normalized ratio [INR] ≥1.5) with encephalopathy in a patient with no prior history of liver disease, with onset of symptoms within 28 days of the inciting event. Patients may have either a history of acetaminophen overdose (defined as >4 g/day within 7 days of presentation) and/or detectable acetaminophen levels in the serum, with a pattern of liver function tests typical for acetaminophen toxicity (bilirubin < 10 mg/dL and alanine aminotransferase (ALT) ≥1000 IU/L), or a diagnosis of hepatitis A, hepatitis B, drug-induced liver injury, autoimmune hepatitis or indeterminate cause based on standard criteria.
3. ALI patients may also be enrolled (those meeting the above criteria plus coagulopathy (INR ≥ 2.0) and no evidence of encephalopathy)
4. Written informed consent from the patient (ALI) or patient's legally authorized representative or family member if he/she is considered encephalopathic (ALF).
5. Ammonia level ≥60 μmol/L at baseline (within 8h prior to T0/initiation of infusion).
6. Serum creatinine levels as follows:

   1. Cohort 1: Creatinine ≤1.5 mg/dL; and
   2. Cohort 2: Creatinine >1.5 mg/dL and <10mg/dL.
7. Mean arterial pressure of >65 mmHg.

Exclusion Criteria:

1. History of chronic liver disease.
2. Signs of overt cerebral herniation, or uncontrolled intracranial hypertension by intracranial pressure (ICP) monitoring (if applicable).
3. Evidence of Wilson's disease, alcoholic hepatitis, biliary obstruction, ischemic hepatitis, severe acute renal tubular necrosis (ATN) due to shock, or any patient with ongoing hypotension.
4. Significant gastrointestinal bleeding (coffee grounds per nasogastric tube and/or melena).
5. Hemodynamic instability, defined by a mean arterial pressure of <65 mmHg.
6. Cardiopulmonary complications such as pulmonary edema, aspiration pneumonia, heart failure.
7. QT interval of >500msec at baseline EKG.
8. Pregnancy.
9. History of malignancy that has not been cured or any cancer in remission for less than 1 within the past 5 year. Non-melanoma skin cancers do not preclude participation in the trial.
10. Concomitant administration of drugs known to interfere with renal excretion of phenylacetylglutamine or those medications that may induce hyperammonemia such as haloperidol, valproic acid and systemic corticosteroids (prohibited during the study). Alternative ammonia modifying agents such as lactulose and rifaximin are not considered standard of care and are prohibited during the study period.
11. Any other health condition that would preclude participation in the study in the judgment of the principal investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-06; Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William M Lee, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (11):
- United States (11):
  - University of California, San Francisco, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - The Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for the overall study will be shared once the study is completed.
Supporting Information: Study Protocol
Time Frame: The public use dataset (PUDS) will be submitted to the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) within six months of the primary outcome publication date. The PUDS will be available through the NIDDK Repository for the period of time required under the NIDDK Data Sharing Policy.
Access Criteria: The STOP-ALF PUDS will be made available without cost to researchers and analysts.

REFERENCES:
- [Background] Lee WM. Etiologies of acute liver failure. Semin Liver Dis. 2008 May;28(2):142-52. doi: 10.1055/s-2008-1073114. PMID 18452114
- [Background] Roberts MS, Angus DC, Bryce CL, Valenta Z, Weissfeld L. Survival after liver transplantation in the United States: a disease-specific analysis of the UNOS database. Liver Transpl. 2004 Jul;10(7):886-97. doi: 10.1002/lt.20137. PMID 15237373
- [Background] Stravitz RT, Kramer DJ. Management of acute liver failure. Nat Rev Gastroenterol Hepatol. 2009 Sep;6(9):542-53. doi: 10.1038/nrgastro.2009.127. Epub 2009 Aug 4. PMID 19652652
- [Background] Blei AT. Pathogenesis of brain edema in fulminant hepatic failure. Prog Liver Dis. 1995;13:311-30. No abstract available. PMID 9224508
- [Background] Jalan R. Pathophysiological basis of therapy of raised intracranial pressure in acute liver failure. Neurochem Int. 2005 Jul;47(1-2):78-83. doi: 10.1016/j.neuint.2005.04.010. PMID 15927306
- [Background] Larsen FS, Wendon J. Prevention and management of brain edema in patients with acute liver failure. Liver Transpl. 2008 Oct;14 Suppl 2:S90-6. doi: 10.1002/lt.21643. PMID 18825686
- [Background] Clemmesen JO, Larsen FS, Kondrup J, Hansen BA, Ott P. Cerebral herniation in patients with acute liver failure is correlated with arterial ammonia concentration. Hepatology. 1999 Mar;29(3):648-53. doi: 10.1002/hep.510290309. PMID 10051463
- [Background] Blei AT, Larsen FS. Pathophysiology of cerebral edema in fulminant hepatic failure. J Hepatol. 1999 Oct;31(4):771-6. doi: 10.1016/s0168-8278(99)80361-4. No abstract available. PMID 10551405
- [Background] Bhatia V, Singh R, Acharya SK. Predictive value of arterial ammonia for complications and outcome in acute liver failure. Gut. 2006 Jan;55(1):98-104. doi: 10.1136/gut.2004.061754. Epub 2005 Jul 15. PMID 16024550
- [Background] Traber PG, Dal Canto M, Ganger DR, Blei AT. Electron microscopic evaluation of brain edema in rabbits with galactosamine-induced fulminant hepatic failure: ultrastructure and integrity of the blood-brain barrier. Hepatology. 1987 Nov-Dec;7(6):1272-7. doi: 10.1002/hep.1840070616. PMID 3679092
- [Background] Cordoba J, Gottstein J, Blei AT. Glutamine, myo-inositol, and organic brain osmolytes after portocaval anastomosis in the rat: implications for ammonia-induced brain edema. Hepatology. 1996 Oct;24(4):919-23. doi: 10.1002/hep.510240427. PMID 8855198
- [Background] Rose C, Michalak A, Rao KV, Quack G, Kircheis G, Butterworth RF. L-ornithine-L-aspartate lowers plasma and cerebrospinal fluid ammonia and prevents brain edema in rats with acute liver failure. Hepatology. 1999 Sep;30(3):636-40. doi: 10.1002/hep.510300311. PMID 10462368
- [Background] Rose C, Michalak A, Pannunzio M, Chatauret N, Rambaldi A, Butterworth RF. Mild hypothermia delays the onset of coma and prevents brain edema and extracellular brain glutamate accumulation in rats with acute liver failure. Hepatology. 2000 Apr;31(4):872-7. doi: 10.1053/he.2000.5923. PMID 10733542
- [Background] Jalan R, Wright G, Davies NA, Hodges SJ. L-Ornithine phenylacetate (OP): a novel treatment for hyperammonemia and hepatic encephalopathy. Med Hypotheses. 2007;69(5):1064-9. doi: 10.1016/j.mehy.2006.12.061. Epub 2007 Apr 27. PMID 17467190
- [Background] Polson J, Lee WM; American Association for the Study of Liver Disease. AASLD position paper: the management of acute liver failure. Hepatology. 2005 May;41(5):1179-97. doi: 10.1002/hep.20703. No abstract available. PMID 15841455
- [Background] Sterling RK, Luketic VA, Sanyal AJ, Shiffman ML. Treatment of fulminant hepatic failure with intravenous prostaglandin E1. Liver Transpl Surg. 1998 Sep;4(5):424-31. doi: 10.1002/lt.500040501. PMID 9724481
- [Background] O'Grady JG, Gimson AE, O'Brien CJ, Pucknell A, Hughes RD, Williams R. Controlled trials of charcoal hemoperfusion and prognostic factors in fulminant hepatic failure. Gastroenterology. 1988 May;94(5 Pt 1):1186-92. doi: 10.1016/0016-5085(88)90011-x. PMID 3280388
- [Background] Jalan R, Olde Damink SW, Deutz NE, Hayes PC, Lee A. Moderate hypothermia in patients with acute liver failure and uncontrolled intracranial hypertension. Gastroenterology. 2004 Nov;127(5):1338-46. doi: 10.1053/j.gastro.2004.08.005. PMID 15521003
- [Background] Stravitz RT, Larsen FS. Therapeutic hypothermia for acute liver failure. Crit Care Med. 2009 Jul;37(7 Suppl):S258-64. doi: 10.1097/CCM.0b013e3181aa5fb8. PMID 19535956
- [Background] Randomised trial of steroid therapy in acute liver failure. Report from the European Association for the Study of the Liver (EASL). Gut. 1979 Jul;20(7):620-3. doi: 10.1136/gut.20.7.620. PMID 385456
- [Background] Kumar M, Satapathy S, Monga R, Das K, Hissar S, Pande C, Sharma BC, Sarin SK. A randomized controlled trial of lamivudine to treat acute hepatitis B. Hepatology. 2007 Jan;45(1):97-101. doi: 10.1002/hep.21486. PMID 17187417
- [Background] Ichai P, Duclos-Vallee JC, Guettier C, Hamida SB, Antonini T, Delvart V, Saliba F, Azoulay D, Castaing D, Samuel D. Usefulness of corticosteroids for the treatment of severe and fulminant forms of autoimmune hepatitis. Liver Transpl. 2007 Jul;13(7):996-1003. doi: 10.1002/lt.21036. PMID 17370335
- [Background] Makin AJ, Wendon J, Williams R. A 7-year experience of severe acetaminophen-induced hepatotoxicity (1987-1993). Gastroenterology. 1995 Dec;109(6):1907-16. doi: 10.1016/0016-5085(95)90758-0. PMID 7498656
- [Background] Larson AM, Polson J, Fontana RJ, Davern TJ, Lalani E, Hynan LS, Reisch JS, Schiodt FV, Ostapowicz G, Shakil AO, Lee WM; Acute Liver Failure Study Group. Acetaminophen-induced acute liver failure: results of a United States multicenter, prospective study. Hepatology. 2005 Dec;42(6):1364-72. doi: 10.1002/hep.20948. PMID 16317692
- [Background] Lee WM, Hynan LS, Rossaro L, Fontana RJ, Stravitz RT, Larson AM, Davern TJ 2nd, Murray NG, McCashland T, Reisch JS, Robuck PR; Acute Liver Failure Study Group. Intravenous N-acetylcysteine improves transplant-free survival in early stage non-acetaminophen acute liver failure. Gastroenterology. 2009 Sep;137(3):856-64, 864.e1. doi: 10.1053/j.gastro.2009.06.006. Epub 2009 Jun 12. PMID 19524577
- [Background] Liou IW, Larson AM. Role of liver transplantation in acute liver failure. Semin Liver Dis. 2008 May;28(2):201-9. doi: 10.1055/s-2008-1073119. PMID 18452119
- [Background] Stravitz RT, Kramer AH, Davern T, Shaikh AO, Caldwell SH, Mehta RL, Blei AT, Fontana RJ, McGuire BM, Rossaro L, Smith AD, Lee WM; Acute Liver Failure Study Group. Intensive care of patients with acute liver failure: recommendations of the U.S. Acute Liver Failure Study Group. Crit Care Med. 2007 Nov;35(11):2498-508. doi: 10.1097/01.CCM.0000287592.94554.5F. PMID 17901832
- [Background] Acharya SK, Bhatia V, Sreenivas V, Khanal S, Panda SK. Efficacy of L-ornithine L-aspartate in acute liver failure: a double-blind, randomized, placebo-controlled study. Gastroenterology. 2009 Jun;136(7):2159-68. doi: 10.1053/j.gastro.2009.02.050. PMID 19505424
- [Background] Jalan R, Lee WM. Treatment of hyperammonemia in liver failure: a tale of two enzymes. Gastroenterology. 2009 Jun;136(7):2048-51. doi: 10.1053/j.gastro.2009.04.016. Epub 2009 May 3. No abstract available. PMID 19409290
- [Background] Davies NA, Wright G, Ytrebo LM, Stadlbauer V, Fuskevag OM, Zwingmann C, Davies DC, Habtesion A, Hodges SJ, Jalan R. L-ornithine and phenylacetate synergistically produce sustained reduction in ammonia and brain water in cirrhotic rats. Hepatology. 2009 Jul;50(1):155-64. doi: 10.1002/hep.22897. PMID 19437490
- [Background] Ytrebo LM, Kristiansen RG, Maehre H, Fuskevag OM, Kalstad T, Revhaug A, Cobos MJ, Jalan R, Rose CF. L-ornithine phenylacetate attenuates increased arterial and extracellular brain ammonia and prevents intracranial hypertension in pigs with acute liver failure. Hepatology. 2009 Jul;50(1):165-74. doi: 10.1002/hep.22917. PMID 19554542
- [Background] Zimmerman L, Jornvall H, Bergstrom J. Phenylacetylglutamine and hippuric acid in uremic and healthy subjects. Nephron. 1990;55(3):265-71. doi: 10.1159/000185973. PMID 2370926
- [Background] Novack, T. (2000). The Orientation Log. The Center for Outcome Measurement in Brain Injury. http://www.tbims.org/combi/olog
- [Derived] Stravitz RT, Fontana RJ, Karvellas C, Durkalski V, McGuire B, Rule JA, Tujios S, Lee WM; Acute Liver Failure Study Group. Future directions in acute liver failure. Hepatology. 2023 Oct 1;78(4):1266-1289. doi: 10.1097/HEP.0000000000000458. Epub 2023 May 16. PMID 37183883
- See also: Acute Liver Failure Study Website — http://www.utsouthwestern.edu/labs/acute-liver/
- See also: Instructional STOP-ALF YouTube Video — http://youtu.be/WUKZWx3Qa7U

RESULTS

PARTICIPANT FLOW:
Groups:
- Maximum Dose Level 3.33 g/24h: Initial infusion of study drug at 0.139 g/h for the first 12 hours (approximately 3.33 g/24h) and maintained at this rate for up to 120 hours.
- Maximum Dose Level 6.65 g/24h: Initial infusion of study drug at a dose of 0.139 g/h for the first 12 hours (approximately 3.33 g/24h); dose increased to 0.277 g/h for the remaining 108 hours (approximately 6.65 g/24h) for a total treatment period of up to 120 hours.
- Maximum Dose Level 10 g/24h: Initial infusion of study drug at a dose of 0.139 g/h for the first 12 hours (approximately 3.33 g/24h); dose increased to 0.277 g/h for the next 12 hours; dose then increased to 0.416 g/h (approximately 10 g/24h) and maintained at this rate for the remaining 96 hours for a total treatment period of up to 120 hours.
- Maximum Dose Level 20g/24h: Study drug infused at a dose of 20g/24h from initiation of infusion for a maximum time of up to 120 hours.
Period: Overall Study
Arm/Group | Maximum Dose Level 3.33 g/24h | Maximum Dose Level 6.65 g/24h | Maximum Dose Level 10 g/24h | Maximum Dose Level 20g/24h
Started | 9 | 10 | 13 | 15
Evaluable (72 Hours on Infusion) | 6 | 6 | 12 | 12
Completed | 9 | 7 | 8 | 10
Not Completed | 0 | 3 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Maximum Dose Level 20g/24h: Study drug infused at a dose of 20g/24h from initiation of infusion for up to 120 hours.
- Total: Total of all reporting groups
Arm/Group | Maximum Dose Level 3.33 g/24h | Maximum Dose Level 6.65 g/24h | Maximum Dose Level 10 g/24h | Maximum Dose Level 20g/24h | Total
Number analyzed (Participants) | 9 | 10 | 13 | 15 | 47
Age, Continuous [Median (Full Range); unit: years] | 32.0 [18.0 to 45.0] | 30.0 [21.1 to 62.0] | 42.0 [26.0 to 64.0] | 35.0 [19.0 to 59.0] | 35.0 [18.0 to 64.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 9 | 11 | 31
  Male | 3 | 5 | 4 | 4 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 5 | 11
  White | 7 | 7 | 8 | 10 | 32
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 10 | 13 | 15 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That do Not Tolerate the Administered Dose and Had Grade 3 or 4 Treatment Emergent Adverse Events as a Measure of Safety and Tolerability
Description: To evaluate the safety and tolerability of OCR-002 in patients with acute liver failure/severe acute liver injury
Time Frame: 30 Days
Population: All patients who consented to the study, completed screening and had the intravenous infusion of study drug initiated
Measure: Count of Participants; unit: Participants
Arm/Group | Maximum Dose Level 3.33 g/24h | Maximum Dose Level 6.65 g/24h | Maximum Dose Level 10 g/24h | Maximum Dose Level 20g/24h
Number analyzed (Participants) | 9 | 10 | 13 | 15
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Measurement of OCR-002 Plasma Concentration
Description: To evaluate the steady state pharmacokinetic and pharmacodynamic profile of OCR-002 in patients with impaired and intact renal function using urinary phenylacetylglutamine (PAGN) as a surrogate marker
Time Frame: 24 Hours after last infusion
Population: All patients who consented to the study and had the intravenous infusion of study drug initiated for up to 120 hours and had results available from serum and urine samples measuring the pharmacokinetic (PK), pharmacodynamic profile (phenylacetic acid (PAA), ornithine) and urinary phenylacetylglutamine (PAGN) levels.
Measure: Mean (Standard Deviation); unit: micrograms per millileter
Arm/Group | Maximum Dose Level 3.33 g/24h | Maximum Dose Level 6.65 g/24h | Maximum Dose Level 10 g/24h | Maximum Dose Level 20g/24h
Number analyzed (Participants) | 8 | 8 | 13 | 15
micrograms per millileter | 65.6 (82.5) | 32.2 (31.4) | 33.4 (24.1) | 104.9 (104.5)

3. Secondary Outcome: Change in Ammonia
Description: To evaluate the effect of OCR-002 on ammonia levels in patients with acute liver failure/severe acute liver injury
Time Frame: Baseline and 72 Hours
Population: All patients who consented to the study and had the intravenous infusion of study drug initiated for up to 72 hours and available venous or arterial ammonia levels.
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- Maximum Dose Level 6.65 g/24h: Initial infusion of study drug at a dose of 0.139 g/h for the first 12 hours (approximately 3.33 g/24h); dose increased to 0.277 g/h for the remaining 108 hours (approximately 6.65 g/24h) for a total treatment period of 120 hours.
- Maximum Dose Level 10 g/24h: Initial infusion of study drug at a dose of 0.139 g/h for the first 12 hours (approximately 3.33 g/24h); dose increased to 0.277 g/h for the next 12 hours; dose then increased to 0.416 g/h (approximately 10 g/24h) and maintained at this rate for the remaining 96 hours for a total treatment period of 120 hours.
- Maximum Dose Level 20g/24h: Study drug infused at a dose of 20g/24h from initiation of infusion for a maximum time of 120 hours.
Arm/Group | Maximum Dose Level 3.33 g/24h | Maximum Dose Level 6.65 g/24h | Maximum Dose Level 10 g/24h | Maximum Dose Level 20g/24h
Number analyzed (Participants) | 6 | 8 | 10 | 12
Percent Change | 41.2 (21.1) | 16.6 (51.4) | 41.8 (35.8) | 38.4 (31.1)

4. Secondary Outcome: Neurological Function Measured by the West Haven Criteria (WHC) for Hepatic Encephalopathy
Description: The West Haven Criteria (WHC) for Hepatic Encephalopathy measures the severity of encephalopathy and patient's level of consciousness. The scale ranges from 0 to 4; a minimum score of 0 represents a better outcome, and a maximum total score of 4 represents a worse outcome. A score of 0 corresponds to normal consciousness and behavior and normal neurological examination. A score of 1 corresponds to mild lack of awareness, shortened attention span, and impaired addition or subtraction; mild asterixis or tremor. A score of 2 corresponds to lethargy, disorientated or inappropriate behavior, obvious asterixis; slurred speech. A score of 3 corresponds to somnolent but arousable, gross disorientation or bizarre behavior, muscle rigidity and clonus; hyperreflexia. A score of 4 corresponds to coma and decerebrate posturing.
Time Frame: 120 hours from start of infusion
Population: All patients who consented to the study and had the intravenous infusion of study drug initiated and West Haven Criteria (WHC) for Hepatic Encephalopathy assessment scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maximum Dose Level 3.33 g/24h | Maximum Dose Level 6.65 g/24h | Maximum Dose Level 10 g/24h | Maximum Dose Level 20g/24h
Number analyzed (Participants) | 5 | 5 | 11 | 13
units on a scale | 2.4 (1.9) | 3.2 (2.0) | 1.6 (1.4) | 1.8 (1.6)

5. Secondary Outcome: Neurological Function Measured by the Orientation Log (O-log)
Description: The orientation log focuses on orientation to place, time, and circumstance. There are 10 items on the orientation log, which are scored 0-3. A spontaneous correct response is awarded 3 points. A spontaneous response that is lacking or incorrect, but a correct response is provided following a logical cue is awarded 2 points. A score of 1 is given if spontaneous and cued responses are lacking or incorrect, but a correct response is provided in a recognition format. A score of 0 is given if the spontaneous, cued, or recognition format does not generate a correct answer. Scores from the 10 items are summed and the final score ranges from 0 to 30.
Time Frame: 30 Days
Population: All patients who consented to the study and had the intravenous infusion of study drug initiated and Orientation log (O-log) assessment scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maximum Dose Level 3.33 g/24h | Maximum Dose Level 6.65 g/24h | Maximum Dose Level 10 g/24h | Maximum Dose Level 20g/24h
Number analyzed (Participants) | 5 | 3 | 6 | 4
units on a scale | 23.8 (0.4) | 24.0 (0.0) | 24.0 (0.0) | 24.0 (0.0)

ADVERSE EVENTS:
Time Frame: Serious adverse events & suspected adverse reactions: Collected from the start of the initial study drug infusion through study completion, i.e., Day 30, death, or withdrawal of consent. Non-serious adverse events: Collected from the start of the initial study drug infusion through 24 hours following the final infusion of study drug (typically Day 5) or for 24 hours following the final infusion of study drug for those patients who do not complete the entire course of study drug administration.
Description: Medical conditions not present prior to the start of the initial study drug infusion but emerge thereafter are reported, including exacerbation of pre-existing medical conditions & clinically significant, treatment-emergent lab abnormalities. A safety follow-up visit is performed 30 days after the start of the initial study drug infusion. An independent site monitor performs data verification to ensure all adverse events (AEs) are reported as defined in the protocol.
Arm/Group | Maximum Dose Level 3.33 g/24h | Maximum Dose Level 6.65 g/24h | Maximum Dose Level 10 g/24h | Maximum Dose Level 20g/24h
All-Cause Mortality (participants affected / at risk) | 2/9 | 3/10 | 2/13 | 4/15
Serious Adverse Events (participants affected / at risk) | 5/9 | 3/10 | 4/13 | 4/15
Other Adverse Events (participants affected / at risk) | 8/9 | 5/10 | 9/13 | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maximum Dose Level 3.33 g/24h (N=9) | Maximum Dose Level 6.65 g/24h (N=10) | Maximum Dose Level 10 g/24h (N=13) | Maximum Dose Level 20g/24h (N=15)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Compartment syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain edema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neurological decompensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maximum Dose Level 3.33 g/24h (N=9) | Maximum Dose Level 6.65 g/24h (N=10) | Maximum Dose Level 10 g/24h (N=13) | Maximum Dose Level 20g/24h (N=15)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alcohol withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT interval (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hepatic encephalopathy (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Oedema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (7) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Red man syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (7) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT01548690/Prot_SAP_000.pdf